CLINICAL TRIAL: NCT05169333
Title: The Oxford Risk Factors And Non-Invasive Imaging Study
Acronym: ORFAN
Status: Recruiting | Type: Observational
Sponsor: University of Oxford (Other)
Collaborators: Caristo Diagnostics Limited (Industry); Oxford University Hospitals NHS Trust (Other); British Heart Foundation (Other); Innovate UK (Other Government); European Commission (Other); National Consortium of Intelligent Medical Imaging (Unknown)
Responsible Party: Sponsor
Other Study IDs: The ORFAN Study
Record Dates: First submitted 2021-10-12; First posted 2021-12-23 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Cardiovascular Diseases; Cardiovascular Risk Factors
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 15 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Group 1: Participants attending cardiology department, hypertension or outpatient clinics.
- Group 2: Participants who are recruited prospectively, during their clinically indicated CT scan, and they are followed-up prospectively for clinical endpoints; A follow-up CCTA at least 6 months later will be offered to a subgroup of these patients, to assess disease progression.
- Group 3: Individuals where at least 6 months have elapsed from previous CCTA will undergo repeat CCTA scan and enter prospective follow up for clinical endpoints.
- Group 4: Cohort of consecutive patients who have undergone clinical CTAs or unenhanced CT chest, abdomen and pelvis in the past, linking the index CT scan with prospective outcomes collection already accumulated.

SUMMARY:
ORFAN is a prospective, multi-centre, multi-ethnic cohort observational study collecting CT scans, biological material and outcomes data, to develop and validate novel biomarkers of cardiometabolic and other disease risk.

DETAILED DESCRIPTION:
The ORFAN registry will include unselected, consecutive patients undergoing CT scans (coronary CT angiograms (CCTA), CT chest, abdomen and pelvis scans) collected at the participating centres. The study will combine imaging data with patient demographics and clinical information (including prospective outcomes) to aid the development and/or validation of new or existing image analysis algorithms and software tools to improve diagnosis, clinical risk discrimination and prediction. Specifically, ORFAN will evaluate the specificity, utility and predictive value of newly developed image analysis methods. ORFAN will recruit and follow-up patients prospectively, linking the index CT scan with blood biomarkers, genetic information as well as information on disease progression (recorded through follow-up CT scans) and clinical outcomes data.

The study will also collect CT scans performed in the past and link them with clinical factors and prospective outcomes data collected after the index scan was performed.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for study Arms 1, 2 and 3:

* Participant is willing and able to give informed consent for participation in the study.
* Male or Female, aged 18 -99 years.

Inclusion Criteria for study Arm 4:

• Male or Female, aged 18 -99 years.

Exclusion Criteria:

Exclusion Criteria for Study Arms 1, 2 and 3:

* Unable or unwilling to consent
* Active cancer

Exclusion Criteria for Study Arm 4:

* Participation in Study Arms 1, 2 or 3
* Existing opt-out from use of data for research purposes

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from secondary and tertiary NHS care providers in the UK and from international sites.
Sampling Method: Non-Probability Sample
Enrollment: 250000 (Estimated)
Dates: Start 2016-02-23 (Actual); Primary Completion 2030-02 (Estimated); Study Completion 2030-02 (Estimated)

PRIMARY OUTCOMES:
Cardiac and all cause mortality | 15 years
  Using novel image analysis methods, clinical risk factors, and blood biomarkers to predict future cardiac and all-cause mortality over a period of 15 years post CT scan.
Non-fatal vascular events | 15 years
  Using novel image analysis methods, clinical risk factors, and blood biomarkers to predict future non-fatal vascular events over a period of 15 years post CT scan.
Cardiac and non-cardiac findings by Computed Tomography | 15 years
  Using novel image analysis methods, clinical risk factors, and blood biomarkers to detect pathology from Computed Tomography images.
Progression of disease | 15 years
  Using novel image analysis methods, clinical risk factors, and blood biomarkers to predict progression of cardiometabolic diseases over a period of 15 years post index CT scan.

SECONDARY OUTCOMES:
Cardiovascular risk factors | 15 years
  Using novel image analysis methods and blood biomarkers, to detect and monitor cardiovascular risk factors and responsiveness to routine clinical care
Hospital admissions for any reason classified using ICD10 | 15 years
  Using novel image analysis methods, to predict hospital admissions over a period of 15 years post CT scan
Genotyping | 15 years
  Using genotyping to predict clinical phenotypes
Progression of cardiovascular disease | 15 years
  Using novel image analysis methods, clinical risk factors, and blood biomarkers to predict disease progression measured by CT scans
Validation and refinement of the CaRi Image analysis platform | 15 years
  Validate the prognostic and diagnostic performance of CaRi Image analysis platform against the other study outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Antoniades, Principal Investigator — University of Oxford
Locations (37):
- United States (3):
  - NIH National Heart, Lunch, and Blood Institute, Bethesda, Maryland
  - Mayo Clinic, Rochester, Minnesota
  - Cleveland Clinic Heart and Vascular Institute, Cleveland, Ohio
- Australia (2):
  - Flinders University, Adelaide
  - The University of Sydney, Sydney
- University Hospitals Leuven, Leuven, Belgium
- China (2):
  - Fudan University, Shanghai
  - TEDA International Cardiovascular Hospital, Tianjin
- Almaviva Sante - Clinique Axium, Aix-en-Provence, France
- Germany (2):
  - Friedrich-Alexander-Universitat Erlangen-Nurmberg, Erlangen
  - University Hospital Ulm, Ulm
- Lefkos Stavros Clinic, Athens, Greece
- MTA-SE Cardiovascular Imaging Research Group, Budapest, Hungary
- Centro Cardiologico Monzino IRCCS, University of Milan, Milan, Italy
- Oita University, Ōita, Japan
- Netherlands (2):
  - Amsterdam Universitair Medische Centra, Amsterdam
  - Zuyderland Medical Centre, Sittard
- University of Medicine and Pharmacy of Targu Mures, Târgu Mureş, Romania
- Seoul National University, Seoul, South Korea
- Cleveland Clinic Abu Dhabi, Abu Dhabi, United Arab Emirates
- United Kingdom (17):
  - Royal United Hospitals Bath NHS Foundation Trust, Bath
  - Sandwell and West Birmingham Hospitals NHS Trust, Birmingham
  - University Hospitals Birmingham NHS Trust, Birmingham
  - Royal Papworth Hospital NHS Trust, Cambridge
  - University of Edinburgh, Royal Infirmary, Edinburgh
  - Golden Jubilee National Hospital, Glasgow
  - NHS Greater Glasgow and Clyde, Glasgow
  - Leeds Teaching Hospitals NHS Trust, Leeds
  - University Hosptials of Leicester NHS Trust, Leicester
  - Liverpool Heart and Chest Hospital, Liverpool
  - Barts Health NHS Trust, London
  - Guy's and St Thomas' NHS Foundation Trust, London
  - Royal Brompton and Harefield Hospitals, London
  - University Hospital of Manchester NHS Foundation Trust, Manchester
  - Milton Keynes University Hospital, Milton Keynes
  - Oxford University Hospitals NHS Foundation Trust, Oxford
  - Heart and Lung Centre, New Cross Hospital, Wolverhampton

REFERENCES:
- [Derived] Westwood M, Armstrong N, Krijkamp E, Perry M, Noake C, Tsiachristas A, Corro-Ramos I. A cloud-based medical device for predicting cardiac risk in suspected coronary artery disease: a rapid review and conceptual economic model. Health Technol Assess. 2024 Jul;28(31):1-105. doi: 10.3310/WYGC4096. PMID 39023142